CLINICAL TRIAL: NCT06107179
Title: Non-invasive Monitoring of Disease Activity in Pediatric Inflammatory Bowel Diseases Using Multispectral Optoacoustic Tomography
Brief Title: Monitoring of Pediatric Inflammatory Bowel Diseases Using Multispectral Optoacoustic Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 23-278-Bm
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: MSOT; Optoacoustics; Photoacoustics
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohns Disease: Patients with Crohns Disease
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography
- Ulcerative Colitis: Patients with Ulcerative Colitis
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography

INTERVENTIONS:
Diagnostic Test: Multispectral Optoacoustic Tomography — In MSOT, laser light is emitted into the target tissue via a handheld probe. Thermoelastic expansion of various molecules in the target area generates ultrasound waves that are detected by the transducer. The detected signals are reconstructed into images using algorithms. Spectral analysis of the optoacoustic signal at different wavelengths in the near-infrared range can detect individual chromophores, such as oxygenated and deoxygenated hemoglobin.

SUMMARY:
In this clinical trial, the intestinal wall of pediatric patients with Crohns disease and Ulcerative Colitis will be assessed with multispectral optoacoustic tomography (MSOT) to characterize the optoacoustic signal of the intestinal wall and to monitor disease activity.

The goal of this clinical trial is to compare the optoacoustic signal in the intestinal wall of children with inflammatory bowel diseases. The main questions it aims to answer are:

* How does the optoacoustic signal in children with inflammatory bowel diseases change over time?
* How does the optoacoustic signal in children with inflammatory bowel diseases change when they receive therapy? Participants will be examined with multispectral optoacoustic tomography.

DETAILED DESCRIPTION:
In this study, the disease activity of children and adolescents with inflammatory bowel disease (IBD) will be assessed non-invasively by multispectral optoacoustic tomography (MSOT). IBDs play an important role in pediatric and adolescent medicine. The most common entities in the IBS group are Crohn's disease (CD) and ulcerative colitis (UC). Patients with CD develop chronic intermittent transmural inflammation of the gastrointestinal (GI) tract. Symptoms include diarrhea, hematochezia, abdominal pain, and malnutrition. Complications of the disease include fistula formation, perforations, and bleeding.The basis for many clinical decisions is the detection of disease activity.There are limitations to previous imaging methods for routine monitoring that are particularly relevant in pediatric and adolescent medicine.The use of contrast media, sedation, and invasive procedures are a burden for pediatric patients*.Multispectral optoacoustic tomography (MSOT) offers a radiation-free and noninvasive alternative for detecting disease activity. Quantitative assessment of hemoglobin signal in the bowel wall of patients with CD could previously be correlated with endoscopically detected disease activity. The aim of this study is to evaluate whether MSOT also allows monitoring of chronic inflammatory diseases in children. For this purpose, children in different stages of disease who regularly receive intravenous therapeutic administrations of biologics (e.g. infliximab) in our hospital will be examined. The investigators think that by means of MSOT different stages and courses of the diseases could be measured non-invasively and thus invasive measures in children could be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Existing diagnosis of CD or UC, or suspected CD or UC at initial diagnosis.
* Age 2 - 18 years
* Written declaration of consent from parents / legal guardians

Exclusion Criteria:

* Pregnancy
* Nursing mothers
* Cardiopulmonary unstable patients*: Need for continuous cardiopulmonary monitoring
* Tattoo in the area of the examination field
* Subcutaneous fat > 3 cm

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: IBD patients will be enrolled from the department of pediatric gastroenterology of the University hospital Erlangen, a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
MSOT signal for hemoglobin in the intestinal wall of participants | 6 - 12 months
  Longitudinal analysis of MSOT signal for oxygenated and deoxygenated hemoglobin in the intestinal wall of children and adolescents with CD and UC.

SECONDARY OUTCOMES:
Quantitative comparison of the signal of oxygenated and deoxygenated hemoglobin measured by MSOT in inflamed and non-inflamed intestinal wall sections of children and adolescents with CD and UC. | 6 - 12 months
  Quantitative comparison of the signal of oxygenated and deoxygenated hemoglobin measured by MSOT in inflamed and non-inflamed intestinal wall sections of children and adolescents with CD and UC.
Quantitative comparison of oxygenated and deoxygenated hemoglobin signal measured by MSOT in different intestinal wall sections of children and adolescents with CD and UC. | 6 - 12 months
  Quantitative comparison of oxygenated and deoxygenated hemoglobin signal measured by MSOT in different intestinal wall sections of children and adolescents with CD and UC.
-Quantitative comparison of the quantitative fraction of fibrosis/collagen signal determined by MSOT in intestinal walls of children with IBD of different entities (CD and UC) | 6 - 12 months
  -Quantitative comparison of the quantitative fraction of fibrosis/collagen signal determined by MSOT in intestinal walls of children with IBD of different entities (CD and UC)
Quantitative amount of single wavelength signal in a.u. | 6 - 12 months
  single wavelength signals in the intestinal wall of children with different entities of IBD (CD vs. UC) derived by MSOT in arbitrary units (a.u.)
Optoacoustic spectrum in a.u | 6 - 12 months
  Optoacoustic spectrum in the intestinal wall of children with different entities of IBD (CD vs. UC) derived by MSOT in arbitrary units (a.u.)
Endoscopic extent of inflammation (if applicable) | 6 - 12 months
  Assessment of inflammation in endoscopies within different entities of IBD (CD vs. UC)
Histological extent of inflammation and fibrosis (if applicable) | 6 - 12 months
  Assessment of inflammation and fibrosis in histological samples from biopsies within different entities of IBD (CD vs. UC)
Clinical evaluation | 6 - 12 months
  Assessement of clinical disease status by PCDAI or PUCAI according to the CED within different entities of IBD (CD vs. UC)
Ultrasound | 6 - 12 months
  Assessment of disease status by ultrasound within different entities of IBD (CD vs. UC)
Laboratory parameters (blood - c-reactive protein (CrP)) (if applicable) | 6 - 12 months
  Assessment of disease status by laboratory parameters (CrP) within different entities of IBD (CD vs. UC)
Laboratory parameters (stool - Calprotectin) (if applicable) | 6 - 12 months
  Assessment of disease status by laboratory parameters (Calprotectin) within different entities of IBD (CD vs. UC)
MRI (if applicable) | 6 - 12 months
  Assessment of disease status by MRI within different entities of IBD (CD vs. UC)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian P Regensburger, Principal Investigator — Childrens Hospital of the University hospital of Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No